CLINICAL TRIAL: NCT03292679
Title: Craniofacial Applications of 3D Printing
Status: Withdrawn | Type: Observational
Why Stopped: There was lack of internal staff support and could not enroll participants.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Arthur Nam, Assistant Professor, University of Maryland, Baltimore
Other Study IDs: HP-00071854
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Facial Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 3D template: Subjects will have custom models of relevant portions of their facial skeleton printed and used as templates for bending and shaping plates for stabilizing the fracture(s).
  Interventions: Procedure: 3D template

INTERVENTIONS:
Procedure: 3D template — A 3D-printed model of relevant portions of the patient's facial skeleton, based on patient's CT scan will be created. This model will be used to bend titanium reconstruction plates that are used to stabilize the facial fracture for subjects in the treatment group.
  Bending of the plates will be performed in the operating room during the patient's surgery. Titanium reconstruction plates are used to stabilize the fracture whether or not the individual is in the study. However, for patients that are in the treatment arm of the study, the plates are bent with the aid of the 3D-printed model as template, rather than by free-hand.

SUMMARY:
3D printing is a technology that allows for physical creation of a 3D model (usually made of plastic) based on computer generated 3D images from CT scans. The 3D images of craniofacial skeleton using computer software are routinely generated and, in turn, these 3D images can be used to create a plastic 3D model using a 3D printer.

Unstable or comminuted facial fractures need to be reduced and rigidly fixated using titanium plates and screws. Bending and shaping of the plates is usually performed by free-hand based on the surgeon's estimation of what best fits the fracture.

Often, bending the titanium plates to the shape of pre-injury skeletal contour is difficult when the bone is fractured into many pieces or is unstable, or when the patient is edentulous (missing several teeth). The process can increase the time spent in surgery and the bent plates may not snugly fit the fracture. For these difficult cases, one option is to use commercially manufactured 3D printed patient-specific models. The patient-specific models provide the benefit of correct shape / form for increased surgical accuracy, and decreased intra-operative time. However these commercial models are manufactured at distant facilities and usually require more than 7 days before delivery. As such, they delay time to surgery and cannot be used for urgent surgery. Additionally, the commercially manufactured implants are expensive, significantly increasing the cost of treatment.

The purpose of this study is to explore whether custom plastic models 3D printed at Shock Trauma Center and used for bending and shaping plates for facial fracture repair can improve results of facial fracture reconstruction.

Our plastic surgery division will design and produce facial bone 3D model of patients (with facial fractures) using an in-house 3D printer, then use the 3D model to contour the hardware pre-op or intra-op at the time of fracture repair. We believe that we can achieve better repair, shorter surgery time, and save hardware cost.

DETAILED DESCRIPTION:
The purpose of this study is to:

1. produce 3D printed craniofacial models of patients with facial fracture, then use the 3D models
2. contour (or pre-bend) the appropriate hardware pre-op that is specific for the patient.

Fracture repair in the operating room entails exposure and reduction of the fracture, followed by contouring the hardware to the correct shape to maintain the fracture reduction. However, in unstable or comminuted fractures or in patients missing several teeth, contouring the plate to the correct shape can be time consuming and, sometimes, the plate shape can be inaccurate. Our hypothesis is that using our own 3D model printed on-site to "pre-bend" plates will save intra-operative time and cost, and achieve superior clinical outcome.

Patients will be enrolled to participate if they meet inclusion and exclusion criteria, and provide informed consent.

Additionally, for study subjects, protected health information such as name, date of birth, medical record number, and demographic information (age, sex, ethnic group), Billing and payment information with medical justification, clinical information related to the procedure and follow-up visits will be handled by research personnel for research purposes.

Otherwise, management of the study subjects will be essentially the same as for patients that are not enrolled in the study. This includes CT scans obtained postoperatively to confirm adequate fracture repair, routine clinic follow-up visits (during post-op week 1, week 4, 3 months, 6 months, and/or 1 year after surgery) and additional follow-up visits as may be deemed necessary based on clinical status.

Prior experience of utilizing on-site 3D printing technology in facial reconstruction surgery is limited. If a patient-specific plate is needed, then the plates must be made by commercial manufacturers which usually takes days to produce, and is therefore not suited to treatment of facial trauma.

Trauma plastic surgery division owns and operates a 3D printer. We have experience with CT image processing and have made 3D models of patients facial skeleton (i.e. midface, mandible) that were used as templates for repairing facial fractures.

Patients with complex facial injuries or defects require reconstruction using hardware to restore facial contour and functional stability. In many complex facial reconstructions, surgeons consult commercial companies for expertise in computer aided design and manufacturing of patient-specific implants. The advantages of undergoing this process include (1) in-depth anatomic analysis, (2) improved design of hardware leading to better surgical outcome, and (3) shortened OR time. The disadvantages include length of time required for the production of patient-specific implant (usually 3 to 7 days), and high cost: for example, a mandible 3D model and associated patient-specific reconstruction plate is >$3000.

Three-dimensional printing is an actively evolving technology, especially in surgery. Design modifications and improvement in extrusion technology have made 3D printing made this process much more affordable and relatively easy. It is now possible for individuals (and surgeons!) to generate these 3D models.

Repair of mandible fractures is especially challenging when the patient is edentulous (missing several or all teeth) for several reasons including the smaller bulk of the edentulous mandible, requiring larger reconstructive plates spanning a bigger section of the jaw. Surgery generally takes longer for these patients when compared with non-edentulous patients. A substantial portion of the lengthiness is due to time spent bending the plate.

The rationale for this IRB proposal is to explore the efficacy of 3D models of the patient's fracture that are printed in house as aids for facial fracture reconstruction. We hypothesize that reconstruction with the aid of the models will require shorter OR time, improve bony fixation, without significant increase in overall cost of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with face CT scans
* Patients with facial fractures
* Patient age 12 years or older

Exclusion Criteria:

* Patients without CT scan
* Patients with facial fractures that do not require rigid fixation using hardware
* Patients with facial fractures that do not have normal contralateral bony structures
* Patient age less than 12 years

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to Shock Trauma Plastic Surgery Division for treatment of facial fractures
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Operative time | 24 hours
  Duration of fracture fixation

CONTACTS AND LOCATIONS:
Locations (1):
- Arthur J Nam, Baltimore, Maryland, United States